CLINICAL TRIAL: NCT05019092
Title: Potential Harms and Benefits of Systematic Screening for Deep Vein Thrombosis in Critically Ill Patients
Brief Title: Systematic Screening for Deep Vein Thrombosis in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ettore Marini (Other)
Responsible Party: Sponsor-Investigator, Ettore Marini, Principal Investigator, University Of Perugia
Organization: University Of Perugia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TVP_UTI_1
Record Dates: First submitted 2021-08-05; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening (Experimental): Ultrasound (US) examination of lower limbs 48 hours after admission and again after 3-5 days (5-7 days after the admission)
  Interventions: Diagnostic Test: Ultrasound examination of lower limb veins
- Control (No Intervention): Ultrasound (US) examination according to the clinical evaluation of risk factors for deep vein thrombosis (DVT) and life-threatening bleeding, based on the standard of care (SOC) of the enrolling institution.

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of lower limb veins — Ultrasound examination will be performed by trained physicians using a commercially available ultrasound system and 5.0-15.0 MHz linear probe. The examinations consists of a comprehensive B-mode ultrasound protocol, from thigh to ankle, employing compression and color-Doppler at selected sites, according to the Consensus Conference of the Society of Radiologists in Ultrasound.
  Arms: Screening

SUMMARY:
Background: venous thromboembolism (VTE) is a common complication in critically ill patients, admitted to the Intensive Care Units (ICUs). At the present time, there is no validated score to estimate risks and benefits of antithrombotic pharmacological prophylaxis in this subset of patients.

Aim of the study: investigating potential harms and benefits of a protocol for systematic screening of DVT in critically ill patients, admitted to an ICU.

Expected relevance: systematic screening for deep vein thrombosis (DVT) through ultrasound (US) lower limb veins examination could help defining the indication to antithrombotic pharmacological treatment, but no protocol of systematic screening has been validated so far. Furthermore, the screening could be associated with over-diagnosis and consequent over-treatment, as well as increased management burden for the caregivers and higher healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Admission to the ICU

Exclusion Criteria:

* duration of stay in ICU <5 days
* SARS-CoV-2 infection
* established DVT or pulmonary embolism at admission
* established coagulation disorder
* presence of inferior vena cava filter at the admission
* admission/discharge to the ICU of another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of deep vein thrombosis | hospitalization in UTI, an average of 10 days
  Diagnosis of deep vein thrombosis

SECONDARY OUTCOMES:
Progression of deep vein thrombosis (DVT) | hospitalization in UTI, an average of 10 days
  Extension of a previously diagnosed DVT to a more proximal site
Prophylaxis/ treatment of venous thromboembolism (VTE) | hospitalization in UTI, an average of 10 days
  Necessity of prophylaxis/ treatment of VTE and its possible modifications during the stay in Intensive Care Unit
Incidence of pulmonary embolism | hospitalization in UTI, an average of 10 days
  Findings of pulmonary embolism at contrast-enhanced CT scan
Occurrence of major bleeding | hospitalization in UTI, an average of 10 days
  According to the definition of the International Society of Thrombosis and Hemostasis
Occurrence of anemia | hospitalization in UTI, an average of 10 days
  Reduction of hemoglobin >2 g/dL without evidence of active bleeding
Duration of ICU stay | hospitalization in UTI, an average of 10 days
  Duration of ICU stay
Risk of death in ICU | hospitalization in UTI, an average of 10 days
  Death
Risk of death within 3 months after hospital discharge | Within 3 months after hospital discharge
  Death
Risk of new hospital admission within 3 months after hospital discharge | Within 3 months after hospital discharge
  New hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Leonella Pasqualini, MD, Principal Investigator — University Of Perugia
Locations (1):
- Medicine Interna, Angiologia e Malattie da arteriosclerosi, Perugia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Authors agree to share IPD after publication of results. Data will be access on request to the corresponding Author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of results
Access Criteria: Available on request, by the corresponding author

REFERENCES:
- [Derived] Tini G, Moriconi A, Ministrini S, Zullo V, Venanzi E, Mondovecchio G, Campanella T, Marini E, Bianchi M, Carbone F, Pirro M, De Robertis E, Pasqualini L. Ultrasound screening for asymptomatic deep vein thrombosis in critically ill patients: a pilot trial. Intern Emerg Med. 2022 Nov;17(8):2269-2277. doi: 10.1007/s11739-022-03085-8. Epub 2022 Aug 31. PMID 36044159